CLINICAL TRIAL: NCT01700959
Title: Melatonin Intervention For Neurocognitive Deficits in the St. Jude Lifetime Cohort
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MIND; P30CA021765 (NIH); NCI-2012-02053 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2012-09-25; First posted 2012-10-04 (Estimated); Results first posted 2018-06-28 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-03

CONDITIONS: Cancer Malignancies
Keywords: Melatonin; Neurocognitive impairment; Sleep disturbance; Childhood cancer survivors
MeSH Terms: conditions — Parasomnias | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Melatonin (Active Comparator): Participants receive 3 mgs of time-release melatonin 1-2 hours prior to bedtime.
  Interventions: Drug: melatonin
- Placebo (Placebo Comparator): Participants receive a placebo identical to the time-release melatonin and are instructed to take it 1-2 hours prior to bedtime.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: melatonin — Melatonin 3mg time release will be given. Participants will be instructed to take one 3mg time released tablet by mouth approximately 1-2 hours before initiating sleep onset, preferably at the same time each night.
  Other Names: N-Acetyl-5-Methoxytryptamine
  Arms: Melatonin
Drug: placebo — Placebo tablets to match the melatonin will be comprised of inert substances.
  Arms: Placebo

SUMMARY:
Primary objective:

1. To examine the efficacy of melatonin treatment on neurocognitive functioning in adult survivors of childhood cancer.

Secondary objectives:

1. To evaluate the efficacy of melatonin treatment on delayed sleep onset latency in long-term childhood cancer survivors.
2. To investigate whether improvement in sleep onset latency due to melatonin treatment is associated with neurocognitive improvement in long-term childhood cancer survivors.

This study is a randomized double-blind placebo controlled trial of time release melatonin for adult survivors of childhood cancer who demonstrate impaired neurocognitive functioning and/or difficulty falling asleep.

DETAILED DESCRIPTION:
All participants undergo a general neurocognitive evaluation at baseline and 6-month follow-up, focused on assessment of intelligence, academic skills, attention, processing speed, memory and executive functions.

Sleep parameters using self-report and actigraphy will be assessed at three time points during the study: Baseline, 3-months, and 6-months.

Participants will be divided into 3 mutually exclusive groups:

* Cohort 1: Participant has neurocognitive impairment defined as performance on at least one measure of attention, memory, and/or executive functioning at or below the 10th percentile, AND is absent of delayed sleep onset latency defined as an inability to fall asleep within 30 minutes less than once a week during the past month.
* Cohort 2: Participant has neurocognitive impairment defined as performance on at least one measure of attention, memory, and/or executive functioning at or below the 10th percentile, AND has delayed sleep onset latency defined as self-report of an inability to fall asleep within 30 minutes at least once a week during the past month.
* Cohort 3: Participant is absent of neurocognitive impairment defined as performance >10th percentile on all six measures of attention, memory, and executive functioning, AND has delayed sleep onset latency defined as self-report of an inability to fall asleep within 30 minutes > once a week during the past month.

Within each group, participants will be randomly assigned to take either 3 mgs of time release melatonin or placebo 1-2 hours before bedtime each night for 6 months.

Psychosocial measures of health-related quality of life and psychological distress will be completed at baseline and following 6 months of melatonin/placebo treatment.

Biological samples for serum melatonin levels will be collected at baseline and at the 6 month follow-up evaluation.

ELIGIBILITY:
Inclusion Criteria:

* A St. Jude Life participant who was previously treated at St. Jude Children's Research Hospital
* 10 or more years from diagnosis
* 18 years of age or older
* Able to speak and understand the English language
* Participant has a full scale intelligence quotient (FSIQ) score >79.
* Cohort 1 participant:

  * Has neurocognitive impairment defined as performance on at least one measure of attention, memory, and/or executive functioning ≤10th percentile.
  * Is absent of delayed sleep onset latency defined as an inability to fall asleep within 30 minutes < once a week during the past month.
* Cohort 2 participant:

  * Has neurocognitive impairment defined as performance on at least one measure of attention, memory, and/or executive functioning ≤10th percentile.
  * Has delayed sleep onset latency defined as self-report of an inability to fall asleep within 30 minutes ≥ once a week during the past month.
* Cohort 3 participant:

  * Is absent of neurocognitive impairment defined as performance >10th percentile on all six measures of attention, memory, and executive functioning.
  * Has delayed sleep onset latency defined as self-report of an inability to fall asleep within 30 minutes ≥ once a week during the past month.
* Female participant of childbearing age must not be pregnant or lactating
* Female research participant of childbearing age and male research participant of child fathering potential agrees to use safe contraceptive methods

Exclusion Criteria:

* Known allergy to melatonin or any ingredients of the study product or placebo
* Participant currently is taking melatonin
* Known sleep apnea or medically treated sleep disorder (e.g. restless leg syndrome)
* Known diabetes mellitus - insulin treated
* Participant has uncontrolled seizure disorder in past 12 months
* Reported current illicit drug or alcohol abuse or dependence
* Reported current major psychiatric illness (i.e. schizophrenia, bipolar disorder)
* Current treatment with: (1) benzodiazepines or other central nervous system depressants, (2) fluvoxamine, (3) anticoagulants (e.g. coumadin), (4) immunosuppressant or corticosteroids, OR (5) nifedipine (Procardia XL(R))
* Employed in a position that requires night work (i.e. 10pm to 6am)
* Females who are pregnant or lactating/nursing
* History of neurologic event (i.e. traumatic brain injury) unrelated to cancer or its treatment
* Sensory impairment (vision, hearing) that prohibits completion of neurocognitive examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 911 (Actual)
Dates: Start 2013-02-06 (Actual); Primary Completion 2017-04-19 (Actual); Study Completion 2017-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tara Brinkman, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 911 participants were enrolled and screened between February 2013 and June 2017. Of the 911, 298 were ineligible and 33 withdrew prior to randomization. 580 were randomized.
Pre-assignment Details: The remaining 580 participants were categorized into three mutually exclusive groups: (1) neurocognitive impairment (NI) without delayed sleep onset latency (DSOL), (2) NI with DSOL, and (3) No NI with DSOL. Participants were then randomized to take melatonin or placebo.
Groups:
- Melatonin: NI Without DSOL; Melatonin: NI With DSOL; Melatonin: No NI With DSOL: Participants receive 3 mgs of time-release melatonin 1-2 hours prior to bedtime for 6 months.
  melatonin: Melatonin 3mg time release will be given. Participants will be instructed to take one 3mg time released tablet by mouth approximately 1-2 hours before initiating sleep onset, preferably at the same time each night.
- Placebo: NI Without DSOL; Placebo: NI With DSOL; Placebo: No NI With DSOL: Participants receive a placebo identical to the time-release melatonin and are instructed to take it 1-2 hours prior to bedtime for 6 months.
  placebo: Placebo tablets to match the melatonin will be comprised of inert substances.
Period: Overall Study
Arm/Group | Melatonin: NI Without DSOL | Placebo: NI Without DSOL | Melatonin: NI With DSOL | Placebo: NI With DSOL | Melatonin: No NI With DSOL | Placebo: No NI With DSOL
Started | 89 | 88 | 105 | 105 | 96 | 97
Completed | 62 | 64 | 65 | 70 | 69 | 72
Not Completed | 27 | 24 | 40 | 35 | 27 | 25
Not completed — Adverse Event | 0 | 1 | 1 | 2 | 0 | 2
Not completed — Withdrawal by Subject | 15 | 9 | 12 | 11 | 8 | 12
Not completed — Ineligible | 2 | 1 | 2 | 0 | 0 | 1
Not completed — Noncompliant | 9 | 9 | 17 | 18 | 15 | 9
Not completed — Side effects | 1 | 4 | 8 | 4 | 4 | 1

BASELINE CHARACTERISTICS:
Population: Analysis based on intent to treat. Include participants who were randomized and completed the 6-month assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Melatonin: NI Without DSOL | Placebo: NI Without DSOL | Melatonin: NI With DSOL | Placebo: NI With DSOL | Melatonin: No NI With DSOL | Placebo: No NI With DSOL | Total
Number analyzed (Participants) | 58 | 58 | 62 | 68 | 66 | 68 | 380
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.8 (9.1) | 36.4 (8.1) | 32.8 (7.8) | 32.4 (9.3) | 35.8 (9.0) | 36.5 (8.2) | 34.46 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 24 | 37 | 39 | 35 | 46 | 207
  Male | 32 | 34 | 25 | 29 | 31 | 22 | 173
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 4 | 1 | 0 | 7
  Not Hispanic or Latino | 55 | 52 | 59 | 61 | 59 | 61 | 347
  Unknown or Not Reported | 3 | 6 | 1 | 3 | 6 | 7 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 5 | 8 | 9 | 1 | 7 | 36
  White | 52 | 53 | 53 | 59 | 62 | 59 | 338
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 3 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Neurocognitive Function as Measured by Performance on Standardized Tests of Attention, Memory, and Executive Function.
Description: Efficacy of melatonin treatment on neurocognitive functioning in adult survivors of childhood cancer (Cohorts 1 and 2 only). The measures were analyzed to compare change in neurocognitive performance from baseline to 6 months between active treatment and placebo groups. The unit of measure is a standardized z-score with a mean of 0 and standard deviation of 1. A higher z-score represents a better outcome.
Time Frame: Baseline and 6 months after start of therapy
Population: Analysis based on intent to treat. Include participants who were randomized and completed the 6-month assessment.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Melatonin: NI Without DSOL | Placebo: NI Without DSOL | Melatonin: NI With DSOL | Placebo: NI With DSOL | Melatonin: No NI With DSOL | Placebo: No NI With DSOL
Number analyzed (Participants) | 58 | 58 | 62 | 68 | 0 | 0
Z-score
  Auditory Attention Difference | 0.35 (1.02) | 0.18 (0.87) | 0.06 (1.11) | 0.37 (0.96) |  |
  Sustained Attention Difference | 0.06 (1.11) | 0.16 (1.30) | 0.24 (1.16) | 0.08 (1.39) |  |
  Working Memory Difference | 0.17 (0.67) | 0.07 (0.82) | 0.03 (0.75) | 0.004 (0.76) |  |
  Long-term Verbal Memory Difference | 0.02 (1.16) | -0.03 (1.04) | -0.13 (0.98) | -0.15 (1.29) |  |
  Cognitive Flexibility | 0.31 (1.22) | 0.31 (1.060) | 0.31 (1.37) | 0.18 (1.19) |  |
  Cognitive Fluency Difference | 0.14 (0.68) | 0.21 (0.74) | 0.16 (0.64) | 0.18 (0.63) |  |

2. Secondary Outcome: Sleep Onset Latency as Measured by Actigraphy and Self-report.
Description: Efficacy of melatonin on delayed sleep onset latency in long-term childhood cancer survivors (Cohorts 2 and 3 only). The measures were analyzed to compare change in sleep onset latency from baseline to 6 months between active treatment and placebo groups.
Time Frame: Baseline and six months after start of therapy
Population: Analysis based on intent to treat. Includes participants who were randomized and completed the 6-month assessment.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Melatonin: NI Without DSOL | Placebo: NI Without DSOL | Melatonin: NI With DSOL | Placebo: NI With DSOL | Melatonin: No NI With DSOL | Placebo: No NI With DSOL
Number analyzed (Participants) | 0 | 0 | 62 | 68 | 66 | 68
minutes
  Sleep onset latency - actigraphy |  |  | 5.66 (29.70) | -10.96 (30.21) | -8.47 (23.95) | 1.95 (39.71)
  Sleet onset latency - self-report |  |  | -20.59 (23.73) | 17.79 (37.19) | -18.14 (27.06) | -29.03 (64.49)

3. Secondary Outcome: Neurocognitive Function as Measured by Performance on Standardized Tests of Attention, Memory, and Executive Function, and Sleep Onset Latency as Measured by Actigraphy and Self-report.
Description: Investigate whether improvement in sleep onset latency due to melatonin treatment is associated with neurocognitive improvement in long-term childhood cancer survivors (Cohort 2). The change in neurocognitive performance from baseline to 6 months will be examined in relation to change in sleep onset latency. The unit of measure is a standardized z-score with a mean of 0 and standard deviation of 1. The unit of measurement is a correlation coefficient (Pearson's R2). The range is from -1.0 to 1.0. A zero indicates no correlation while values closer to -1.0 or 1.0 reflect a stronger association. A negative correlation suggests that as sleep latency decreased, neurocognitive functioning improved.
Time Frame: Baseline and six months after start of therapy
Population: Analysis based on intent to treat includes Cohort 2 participants randomized to melatonin who completed the 6-month assessment. Cohorts 1 and 3 were not assessed. 2 assessments of the primary outcome collected in Cohort 2 included self-report and actigraphy. 50 is the total number with actigraphy data. Data were missing for 12 participants.
Measure: Number; unit: Z-score
Groups:
- Melatonin: NI With DSOL (Actigraphy): Data by participant actigraphy. Participants receive 3 mgs of time-release melatonin 1-2 hours prior to bedtime for 6 months.
  melatonin: Melatonin 3mg time release will be given. Participants will be instructed to take one 3mg time released tablet by mouth approximately 1-2 hours before initiating sleep onset, preferably at the same time each night.
- Melatonin: NI With DSOL (Self-report): Data by participant self-report. Participants receive 3 mgs of time-release melatonin 1-2 hours prior to bedtime for 6 months.
  melatonin: Melatonin 3mg time release will be given. Participants will be instructed to take one 3mg time released tablet by mouth approximately 1-2 hours before initiating sleep onset, preferably at the same time each night.
Arm/Group | Melatonin: NI With DSOL (Actigraphy) | Melatonin: NI With DSOL (Self-report)
Number analyzed (Participants) | 50 | 62
Z-score
  Auditory Attention Difference | 0.22 | -0.09
  Sustained Attention Difference | -0.10 | -0.16
  Working Memory Difference | 0.04 | -0.001
  Long-term Verbal Memory Difference | 0.07 | -0.02
  Cognitive Flexibility | 0.30 | 0.15
  Cognitive Fluency Difference | -0.22 | 0.03

ADVERSE EVENTS:
Time Frame: Participants were contacted at the end of the first week on study drug then biweekly for the duration of the study, up to 7 months later. Adverse event information was collected by participant reporting and direct questioning.
Arm/Group | Melatonin: NI Without DSOL | Placebo: NI Without DSOL | Melatonin: NI With DSOL | Placebo: NI With DSOL | Melatonin: No NI With DSOL | Placebo: No NI With DSOL
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/58 | 0/62 | 0/68 | 0/66 | 0/68
Serious Adverse Events (participants affected / at risk) | 2/58 | 2/58 | 9/62 | 6/68 | 2/66 | 10/68
Other Adverse Events (participants affected / at risk) | 37/58 | 37/58 | 52/62 | 60/68 | 57/66 | 58/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Melatonin: NI Without DSOL (N=58) | Placebo: NI Without DSOL (N=58) | Melatonin: NI With DSOL (N=62) | Placebo: NI With DSOL (N=68) | Melatonin: No NI With DSOL (N=66) | Placebo: No NI With DSOL (N=68)
Chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Esophageal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Gallstones (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Trabecular cancer in lungs (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Parotid tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 3 (4)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Concentration impairment (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Kidney infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder perforation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flu-like symptoms (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Maculo-papular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Esophageal dilation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Melatonin: NI Without DSOL (N=58) | Placebo: NI Without DSOL (N=58) | Melatonin: NI With DSOL (N=62) | Placebo: NI With DSOL (N=68) | Melatonin: No NI With DSOL (N=66) | Placebo: No NI With DSOL (N=68)
Palpitation (Cardiac disorders) | 0 (0) | 3 (3) | 2 (2) | 3 (3) | 2 (2) | 6 (10)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 8 (10) | 3 (3) | 10 (10)
Chest pain (Cardiac disorders) | 4 (4) | 2 (2) | 3 (3) | 5 (5) | 4 (4) | 3 (3)
Tinnitus (Ear and labyrinth disorders) | 4 (4) | 7 (7) | 2 (2) | 6 (6) | 3 (4) | 5 (5)
Blurred vision (Eye disorders) | 1 (1) | 3 (4) | 2 (2) | 2 (2) | 6 (6) | 8 (9)
Constipation (Gastrointestinal disorders) | 4 (4) | 3 (3) | 10 (12) | 9 (9) | 6 (6) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 7 (9) | 7 (8) | 10 (14) | 11 (13) | 14 (25) | 17 (20)
Nausea (Gastrointestinal disorders) | 2 (2) | 8 (8) | 4 (5) | 7 (7) | 7 (8) | 13 (15)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Dry mouth (General disorders) | 6 (7) | 6 (6) | 9 (9) | 10 (12) | 9 (11) | 11 (12)
Fatigue (General disorders) | 10 (11) | 13 (20) | 21 (26) | 25 (27) | 21 (23) | 29 (37)
Malaise (General disorders) | 1 (1) | 3 (3) | 5 (5) | 2 (2) | 3 (4) | 7 (7)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 2 (2) | 3 (3)
Dizziness (Nervous system disorders) | 6 (6) | 6 (9) | 16 (20) | 10 (12) | 12 (12) | 12 (14)
Headache (Nervous system disorders) | 15 (20) | 18 (27) | 23 (32) | 27 (32) | 26 (37) | 27 (35)
Hypersomnia (Nervous system disorders) | 6 (8) | 2 (2) | 12 (12) | 12 (14) | 8 (9) | 8 (9)
Nightmares (Nervous system disorders) | 1 (1) | 5 (6) | 3 (3) | 6 (6) | 6 (6) | 8 (11)
Pain (Nervous system disorders) | 3 (3) | 2 (2) | 2 (2) | 4 (4) | 2 (2) | 3 (3)
Somnolence (Nervous system disorders) | 19 (21) | 15 (18) | 23 (24) | 21 (25) | 25 (34) | 29 (36)
Anxiety (Psychiatric disorders) | 5 (5) | 6 (9) | 10 (12) | 11 (17) | 10 (11) | 20 (21)
Delayed orgasm (Psychiatric disorders) | 3 (3) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 4 (4)
Incomnia (Psychiatric disorders) | 11 (16) | 11 (14) | 14 (15) | 20 (21) | 26 (38) | 24 (35)
Libido decreased (Psychiatric disorders) | 3 (3) | 5 (5) | 2 (2) | 2 (2) | 5 (5) | 9 (9)
Restlessness (Psychiatric disorders) | 4 (4) | 6 (8) | 7 (7) | 11 (11) | 9 (10) | 12 (13)
Urinary frequency (Renal and urinary disorders) | 7 (7) | 6 (6) | 9 (9) | 9 (9) | 7 (7) | 6 (6)
Erectile dysfunction (Reproductive system and breast disorders) | 2 (2) | 3 (4) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Irregular menstruation (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 4 (4) | 6 (6) | 5 (5) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (8) | 8 (11) | 12 (13) | 10 (10) | 8 (8) | 11 (11)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3) | 6 (7) | 2 (2) | 6 (6) | 3 (3) | 5 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (9) | 7 (8) | 6 (7) | 10 (10) | 10 (11) | 9 (11)
Maculo=papular rash (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3) | 2 (2) | 8 (9) | 6 (7) | 4 (4)
Concentration impairment (Psychiatric disorders) | 2 (2) | 4 (6) | 9 (9) | 14 (17) | 5 (5) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-11): https://cdn.clinicaltrials.gov/large-docs/59/NCT01700959/Prot_SAP_000.pdf